CLINICAL TRIAL: NCT02827604
Title: Präoperative Und Intraoperative Sonografische Beurteilung Des Unteren Uterinsegmentes im Rahmen Der Re-Sectio Caesarea - Eine Ultraschall- Methoden-Vergleichsstudie
Brief Title: Preoperative and Intraoperative Sonographic Assessment of Lower Uterine Segment Thickness at Term in Women With Previous Cesarean Delivery - a Ultrasound Method Comparison Study
Acronym: SALUTARY
Status: Completed | Type: Observational
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Responsible Party: Principal Investigator, Gregor Seliger, Dr. med., chief resident, Martin-Luther-Universität Halle-Wittenberg
Other Study IDs: SALUTARY
Record Dates: First submitted 2016-07-02; First posted 2016-07-11 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Scar; Previous Cesarean Section
Keywords: Caesarean section; lower uterine segment; sonography
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This prospective, clinical, observational study compares preoperative and intraoperative sonographic assessment of lower uterine segment of women who underwent ≥ second cesarean section.

It is the purpose of the study to assess transabdominal (linear/convex ultrasound probe) and transvaginal approach versus intraoperative sonographic assessment of lower uterine segment.

DETAILED DESCRIPTION:
In 1991, 126.297 (15.3%) women delivered by caesarean section in Germany. Since then, the rate of caesarean section increased steadily over the next 20 years, reaching up to 32.2% in 2011 [https://www.destatis.de]. The absolute risk of uterine rupture in vaginal birth after Caesarean section is 1 in 100 deliveries. The risk of perinatal death or the outcome of extremely neurological impairment is 1 in 1000 deliveries [Cunningham et al., 2009].

Statistically more than 300 pregnant women with a prior caesarean delivery visit daily ultrasound departments of german hospitals to investigate the C-section scar before delivery. They have one important question: Is it possible to predict successful trial of labor after cesarean delivery? [AQUA-Institut] The information for the risk of uterine rupture remains insufficient based only on ultrasonography assessment [Varner et al., 2012].

The measurement technique for lower uterine segment (myometrial) thicknesses in the third trimester have been described by several authors. Using a combination of preoperative transvaginal and transabdominal (linear/convex probe) ultrasound, we compare with intraoperative sonographic assessment of lower uterine segment of women who underwent ≥ second cesarean section.

The aim of the present study is to assess transabdominal (linear/convex ultrasound probe) and transvaginal approach versus intraoperative sonographic assessment of lower uterine segment.

This will allow the investigators to draw conclusions regarding the best method to assessment of lower uterine segment (myometrial) thickness in the third trimester to predict successful trial of labor after cesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

* pregnancy after previous cesarean section
* pregnancy between 37 0/7 and 42 0/7 weeks of gestation
* primary or secondary indication for cesarean section
* ability to give informed consent in german or english

Exclusion Criteria:

* emergency caesarean section
* <18 years old

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with pregnancies after previous cesarean section who referre to the tertiary referral care center.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Difference between preoperative and intraoperative sonographic assessment of lower uterine segment I | intraoperative - just bevore the uterotomy
  Bland-Altman-Plot (mean versus difference) of Method A) Preoperative measurement of minimum myometrium-only thickness overlying the amniotic cavity at the level of the lower uterine segment scar - measured with transabdominal (linear ultrasound probe) and with transvaginal sonography (vaginal ultrasound probe) with the lowest value (thinnest area) being retained AND Method B) Intraoperative measurement of minimum myometrium-only thickness overlying the amniotic cavity at the level of the lower uterine segment scar - measured with intraoperative sonography after preparation of lower uterine segment (linear ultrasound probe)

SECONDARY OUTCOMES:
Difference between preoperative and intraoperative sonographic assessment of lower uterine segment IIA | intraoperative - just bevore the uterotomy
  Bland-Altman-Plot (mean versus difference) of Method A) Preoperative measurement of minimum myometrium-only thickness overlying the amniotic cavity at the level of the lower uterine segment scar - measured with transabdominal (linear ultrasound probe) AND Method B) Intraoperative measurement of minimum myometrium-only thickness overlying the amniotic cavity at the level of the lower uterine segment scar - measured with intraoperative sonography after preparation of lower uterine segment (linear ultrasound probe)
Difference between preoperative and intraoperative sonographic assessment of lower uterine segment IIB | intraoperative - just bevore the uterotomy
  Bland-Altman-Plot (mean versus difference) of Method A) Preoperative measurement of minimum myometrium-only thickness overlying the amniotic cavity at the level of the lower uterine segment scar - measured with transabdominal (convex ultrasound probe) AND Method B) Intraoperative measurement of minimum myometrium-only thickness overlying the amniotic cavity at the level of the lower uterine segment scar - measured with intraoperative sonography after preparation of lower uterine segment (linear ultrasound probe)
Difference between preoperative and intraoperative sonographic assessment of lower uterine segment IIC | intraoperative - just bevore the uterotomy
  Bland-Altman-Plot (mean versus difference) of Method A) Preoperative measurement of minimum myometrium-only thickness overlying the amniotic cavity at the level of the lower uterine segment scar - measured with transvaginal sonography (vaginal ultrasound probe) AND Method B) Intraoperative measurement of minimum myometrium-only thickness overlying the amniotic cavity at the level of the lower uterine segment scar - measured with intraoperative sonography after preparation of lower uterine segment (linear ultrasound probe)

CONTACTS AND LOCATIONS:
Overall Officials: Gregor Seliger, MD, Principal Investigator — Maternity Clinic/Perinatal Treatment Center, Halle university hospital, Martin-Luther-Universität Halle-Wittenberg; Michael Tchirikov, MD, Study Chair — Maternity Clinic/Perinatal Treatment Center, Halle university hospital, Martin-Luther-Universität Halle-Wittenberg
Locations (1):
- Maternity Clinic/Perinatal Treatment Center, Halle university hospital, Martin-Luther-Universität Halle-Wittenberg, Halle, Saxony-Anhalt, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Seliger G, Chaoui K, Lautenschlager C, Riemer M, Tchirikov M. Technique of sonographic assessment of lower uterine segment in women with previous cesarean delivery: a prospective, pre/intraoperative comparative ultrasound study. Arch Gynecol Obstet. 2018 Aug;298(2):297-306. doi: 10.1007/s00404-018-4805-6. Epub 2018 Jun 8. PMID 29948165